CLINICAL TRIAL: NCT00069797
Title: Epidemiology of Coronary Heart Disease in Men Aged 40 and Over
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1233; R01HL068200-05 (NIH)
Record Dates: First submitted 2003-10-01; First posted 2003-10-06 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Atherosclerosis; Coronary Arteriosclerosis; Coronary Disease; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Coronary Disease; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples (serum and plasma), buffy coat for DNA

SUMMARY:
To examine whether the prevalence of subclinical coronary and aortic atherosclerotic disease is different among Japanese in Japan, Japanese in Hawaii, and black and white Americans.

DETAILED DESCRIPTION:
BACKGROUND:

Substantial change toward a more Westernized lifestyle has taken place among younger individuals who were born after World War II (WWII) in non-Western countries including Japan. Data from national sample surveys in Japan clearly demonstrate that risk factor profiles for coronary heart disease (CHD) are very similar to those in the United States (US) in this post WWII cohort. Men in Japan do have a considerably higher prevalence of cigarette smoking and men in the US have a higher prevalence of obesity. CHD mortality among men in Japan is, however, still less than a half of that in the US. Careful review of mortality statistics confirms this. This difference remains unique among industrialized countries.

DESIGN NARRATIVE:

The study is a collaboration between Dr. Akira Sekikawa at the University of Pittsburgh and Dr. J. David Curb of the Pacific Health Research Institute in Honolulu, Hawaii. The study tests the null hypothesis that there are no differences in the extent of atherosclerosis among Japanese men in Japan, Japanese American men in Hawaii, and US white and black men in this post WWII birth cohort. The project is based on recent and ongoing successful Japan/US collaborations in the INTERMAP, INTERLIPID and Honolulu Heart Program studies including development of the first standardized US/Japan diet tables. The investigators will examine 300 white men and 100 black men aged 40-49, randomly selected from Allegheny County, PA, 300 Japanese American men aged 40-49 from the population-based sample recruited from the offspring of the members of the Honolulu Heart Program cohort, and 300 Japanese men aged 40-49, randomly selected from Kusatsu City, Japan. The Japanese recruitment and examination has already been supported in Japan. The extent of atherosclerosis and risk factor profiles for CHD will be evaluated and compared, as well as the relationship of specific risk factors to the measures of atherosclerosis. The measures of subclinical disease proposed include calcium scores of coronary artery and aorta measured by electron beam computed tomography (EBCT) and carotid intima thickness measured by ultrasound. Other proposed measures include dietary intake by food frequency questionnaire, total cholesterol, LDLc, HDLc, lipids by NMR spectroscopy, blood pressure, cigarette smoking, thiocyanate, omega-3 fatty acid, alcohol consumption, body mass index (BMI), intra-abdominal fat, and others.

ELIGIBILITY:
Inclusion:

- Men aged 40-49 at the time of enrollment

Exclusion:

-Individuals with clinical cardiovascular disease (coronary heart disease, stroke), and other severe disease

Ages: 40 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male community members from geographically defined areas (Pittsburgh, PA, Honolulu, HI, and Japan)
Sampling Method: Probability Sample
Enrollment: 1027 (Actual)
Dates: Start 2003-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Intima-media thickness of the carotid artery as well as coronary artery calcification | first visit

CONTACTS AND LOCATIONS:
Overall Officials: J. David Curb, MD, MPH, Principal Investigator — Pacific Health Research Institute; Akira Sekikawa, MD, PhD, PhD, Principal Investigator — University of Pittsburgh; Hirotsugu Ueshima, MD, PhD, Principal Investigator — Shiga University of Medical Science, Japan
Locations (1):
- 130 North Bellefield Avenue, Suite 546, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Sekikawa A, Okamura T, Kadowaki T, Mitsunami K, Murata K, Kashiwagi A, Nakamura Y, Kanda H, Edmundowicz D, Sutton-Tyrrell K, Curb JD, Kuller LH, Ueshima H. [Electron-beam computed tomography for identification of high-risk persons in primary prevention of coronary heart disease in the United States and its implication for Japan]. Nihon Koshu Eisei Zasshi. 2003 Mar;50(3):183-93. Japanese. PMID 12704831
- [Background] Sekikawa A, Horiuchi BY, Edmundowicz D, Ueshima H, Curb JD, Sutton-Tyrrell K, Okamura T, Kadowaki T, Kashiwagi A, Mitsunami K, Murata K, Nakamura Y, Rodriguez BL, Kuller LH. A "natural experiment" in cardiovascular epidemiology in the early 21st century. Heart. 2003 Mar;89(3):255-7. doi: 10.1136/heart.89.3.255. PMID 12591821
- [Result] Sekikawa A, Ueshima H, Zaky WR, Kadowaki T, Edmundowicz D, Okamura T, Sutton-Tyrrell K, Nakamura Y, Egawa K, Kanda H, Kashiwagi A, Kita Y, Maegawa H, Mitsunami K, Murata K, Nishio Y, Tamaki S, Ueno Y, Kuller LH. Much lower prevalence of coronary calcium detected by electron-beam computed tomography among men aged 40-49 in Japan than in the US, despite a less favorable profile of major risk factors. Int J Epidemiol. 2005 Feb;34(1):173-9. doi: 10.1093/ije/dyh285. Epub 2004 Nov 24. PMID 15563587
- [Result] Takamiya T, Kadowaki T, Zaky WR, Ueshima H, Evans RW, Okamura T, Kashiwagi A, Nakamura Y, Kita Y, Tracy RP, Kuller LH, Sekikawa A. The determinants of plasma plasminogen activator inhibitor-1 levels differ for American and Japanese men aged 40-49. Diabetes Res Clin Pract. 2006 May;72(2):176-82. doi: 10.1016/j.diabres.2005.10.015. Epub 2005 Dec 1. PMID 16325297
- [Result] Kadowaki T, Sekikawa A, Murata K, Maegawa H, Takamiya T, Okamura T, El-Saed A, Miyamatsu N, Edmundowicz D, Kita Y, Sutton-Tyrrell K, Kuller LH, Ueshima H. Japanese men have larger areas of visceral adipose tissue than Caucasian men in the same levels of waist circumference in a population-based study. Int J Obes (Lond). 2006 Jul;30(7):1163-5. doi: 10.1038/sj.ijo.0803248. Epub 2006 Jan 31. PMID 16446744
- [Result] Kadowaki T, Sekikawa A, Okamura T, Takamiya T, Kashiwagi A, Zaky WR, Maegawa H, El-Saed A, Nakamura Y, Evans RW, Edmundowicz D, Kita Y, Kuller LH, Ueshima H. Higher levels of adiponectin in American than in Japanese men despite obesity. Metabolism. 2006 Dec;55(12):1561-3. doi: 10.1016/j.metabol.2006.08.004. PMID 17142124
- [Result] Okamura T, Kadowaki T, Sekikawa A, Murata K, Miyamatsu N, Nakamura Y, El-Saed A, Kashiwagi A, Maegawa H, Nishio Y, Takamiya T, Kanda H, Mitsunami K, Kita Y, Edmundowicz D, Tamaki S, Tsujita Y, Kuller LH, Ueshima H. Alcohol consumption and coronary artery calcium in middle-aged Japanese men. Am J Cardiol. 2006 Jul 15;98(2):141-4. doi: 10.1016/j.amjcard.2006.01.095. Epub 2006 May 19. PMID 16828581
- [Result] Abbott RD, Ueshima H, Rodriguez BL, Kadowaki T, Masaki KH, Willcox BJ, Sekikawa A, Kuller LH, Edmundowicz D, Shin C, Kashiwagi A, Nakamura Y, El-Saed A, Okamura T, White R, Curb JD. Coronary artery calcification in Japanese men in Japan and Hawaii. Am J Epidemiol. 2007 Dec 1;166(11):1280-7. doi: 10.1093/aje/kwm201. Epub 2007 Aug 28. PMID 17728270
- [Result] Nakamura Y, Ueno Y, Tamaki S, Kadowaki T, Okamura T, Kita Y, Miyamatsu N, Sekikawa A, Takamiya T, El-Saed A, Sutton-Tyrrell K, Ueshima H. Fish consumption and early atherosclerosis in middle-aged men. Metabolism. 2007 Aug;56(8):1060-4. doi: 10.1016/j.metabol.2007.03.014. PMID 17618950
- [Result] Matsunaga-Irie S, Ueshima H, Zaky WR, Kadowaki T, Evans RW, Okamura T, Takamiya T, Kita Y, Kuller LH, Sekikawa A. Serum ghrelin levels are higher in Caucasian men than Japanese men aged 40-49 years. Diabetes Obes Metab. 2007 Jul;9(4):591-3. doi: 10.1111/j.1463-1326.2006.00627.x. PMID 17587401
- [Result] El-Saed A, Sekikawa A, Edmundowicz D, Evans RW, Sutton-Tyrrell K, Kadowaki T, Choo J, Takamiya T, Kuller LH. Coronary calcification is more predictive of carotid intimal medial thickness in black compared to white middle aged men. Atherosclerosis. 2008 Feb;196(2):913-8. doi: 10.1016/j.atherosclerosis.2007.02.009. Epub 2007 Mar 9. PMID 17350026
- [Result] Sekikawa A, Ueshima H, Sutton-Tyrrell K, Kadowaki T, El-Saed A, Okamura T, Takamiya T, Ueno Y, Evans RW, Nakamura Y, Edmundowicz D, Kashiwagi A, Maegawa H, Kuller LH. Intima-media thickness of the carotid artery and the distribution of lipoprotein subclasses in men aged 40 to 49 years between whites in the United States and the Japanese in Japan for the ERA JUMP study. Metabolism. 2008 Feb;57(2):177-82. doi: 10.1016/j.metabol.2007.08.022. PMID 18191046
- [Result] El-Saed A, Sekikawa A, Zaky RW, Kadowaki T, Takamiya T, Okamura T, Edmundowicz D, Kita Y, Kuller LH, Ueshima H. Association of lipoprotein-associated phospholipase A2 with coronary calcification among American and Japanese men. J Epidemiol. 2007 Nov;17(6):179-85. doi: 10.2188/jea.17.179. PMID 18094516
- [Result] Choo J, Ueshima H, Jang Y, Sutton-Tyrrell K, El-Saed A, Kadowaki T, Takamiya T, Okamura T, Ueno Y, Nakamura Y, Sekikawa A, Curb JD, Kuller LH, Shin C. Difference in carotid intima-media thickness between Korean and Japanese men. Ann Epidemiol. 2008 Apr;18(4):310-5. doi: 10.1016/j.annepidem.2007.08.002. Epub 2007 Nov 5. PMID 17983767
- [Derived] Choo J, Ueshima H, Curb JD, Shin C, Evans RW, El-Saed A, Kadowaki T, Okamura T, Nakata K, Otake T, Miura K, Abbott RD, Sutton-Tyrrell K, Edmundowicz D, Kuller LH, Sekikawa A; ERA-JUMP Study Group. Serum n-6 fatty acids and lipoprotein subclasses in middle-aged men: the population-based cross-sectional ERA-JUMP study. Am J Clin Nutr. 2010 May;91(5):1195-203. doi: 10.3945/ajcn.2009.28500. Epub 2010 Mar 31. PMID 20357040